CLINICAL TRIAL: NCT00213538
Title: Gene Expression Profiling in PBMCs as a Tool for Prediction of Anakinra Responsiveness in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2003/020/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Response to anakinra associated with methotrexate

SUMMARY:
The objective of the study is to identify and validate predictive markers of anakinra responsiveness in RA patients by a transcriptomic approach.

Patients with active RA (ACR criteria) were given subcutaneous anakinra (100mg/d) 3 associated with metotrexate. Anakinra efficacy was evaluated at week 12, using the EULAR response criteria.

A blood sample was collected just before the onset of anakinra treatment and total RNAs were extracted from the peripheral blood mononuclear cells. The [33P] radiolabeled mRNAs were hybridized (duplicate or triplicate) over a set of 10.000 human cDNA probes spotted at a high density on nylon membranes. Data were normalized and filtered to allow the comparison between RNA samples. Statistical analyses were performed with the R software and hierarchical clustering was performed with the Cluster and Tree View softwares.

ELIGIBILITY:
Inclusion Criteria:

* Is age 18 years old or older Satisfies the 1987 American College of Rheumatology revised criteria for Rheumatoid arthritis Has active disease at the time of randomization as indicated by a DAS28> 5.1 Has a disease at least refractory to DMARDs whose methotrexate or leflunomide Is capable of understanding and signing an informed consent form Agrees to use a medically accepted form of contraception during the study

Exclusion Criteria:

* Is pregnant or breast-feeding or without contraception Has significant concurrent medical diseases including cancer or a history of cancer within 5 years of entering the study, uncompensated congestive heart failure, significant active infection or any underlying diseases that could predispose subjects to infections (whose tuberculosis) Has renal disease (creatinin clearance level < 30 ml/min) Has allergy to anakinra Has leukopenia (white blood cells < 1.5 x 109 /l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who Satisfied the 1987 American College of Rheumatology revised criteria for Rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2003-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Auto-antibody level | One year

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Le Loët, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU de rouen - Hôpitaux de Rouen, Rouen, France

REFERENCES:
- [Derived] Bansard C, Lequerre T, Derambure C, Vittecoq O, Hiron M, Daragon A, Pouplin S, Daveau M, Boyer O, Tron F, Le Loet X, Salier JP. Gene profiling predicts rheumatoid arthritis responsiveness to IL-1Ra (anakinra). Rheumatology (Oxford). 2011 Feb;50(2):283-92. doi: 10.1093/rheumatology/keq344. Epub 2010 Nov 8. PMID 21059672